CLINICAL TRIAL: NCT05550766
Title: Prognostic Value of RXR-α in Cutaneous Squamous and Basal Cell Carcinoma: An Immunohistochemical Study.
Brief Title: Prognostic Value of RXR-α in Cutaneous Squamous and Basal Cell Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Fatma Mohammed Hamdan, demonstrator at pathology department, Sohag University
Other Study IDs: Soh-Med-22-09-05
Record Dates: First submitted 2022-09-20; First posted 2022-09-22 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Non-melanoma Skin Cancer

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Vitamin D has a crucial role in cancer control and prevention.vitamin D receptor (VDR) and its heterodimer Retinoid X receptor (RXR) are equally important in the cell. This ligand (vitamin D) and receptors (VDR-RXR) complex together triggers downstream DNA damage response in the cell.

Retinoid receptors are a superfamily of nuclear receptors. The preferred receptor that attaches to VDR is RXR, with its subunits α, β and γ. RXR α is more frequent in the skin than other tissues, while β occurs in internal organs and γ is frequently related to neural disorders.

the investigator hopes to assess prognosis of SCC & BCC by using RXR-α biomarker & attempts to use it in the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Squamous cell carcinoma and basal cell carcinoma.
2. Incisional & excisional biopsies.
3. All the studied cases include sufficient materials for the immunohistochemical study 4. Complete clinical data

Exclusion Criteria:

1. Patients with a history of preoperative chemotherapy and/or radiotherapy.
2. Insufficient or tiny tissue biopsies.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Blocks obtained from cutaneous basal and squamous cell carcinoma tissue from 50 patients.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Prognostic Value of RXR-α in Cutaneous Squamous and Basal Cell Carcinoma | One or two days after staining sections with the marker.
  immuohistochemical expression of RXR-α in Squamous and Basal Cell Carcinoma

IPD SHARING:
Plan to Share IPD: Undecided